CLINICAL TRIAL: NCT04180696
Title: Mid-Q Response Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry); Medtronic Japan Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT18037
Record Dates: First submitted 2019-11-18; First posted 2019-11-27 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Left Bundle-Branch Block; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized after baseline assessment and implant of a CRT system containing the aCRT algorithm. Randomization will be done in a 1:1 ratio to either treatment (aCRT ON, Adaptive Bi-V and LV) or control (aCRT OFF, Nonadaptive CRT) groups. All subjects, independent of randomization assignment, will have a CRT system.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AdaptivCRT ON (aCRT ON, treatment group) (Experimental): AdaptivCRT programmed to "Adaptive Bi-V and LV The aCRT algorithm has been developed to provide RV-synchronized LV pacing when intrinsic AV conduction is normal or BiV pacing otherwise.
  Interventions: Device: aCRT ON
- AdaptivCRT OFF (aCRT OFF, control group) (Active Comparator): AdaptivCRT programmed to "Nonadaptive CRT" (standard CRT). Control group subjects will be optimized per physician's discretion. The method of AV and VV optimization in the control group will be collected.
  Interventions: Device: aCRT OFF

INTERVENTIONS:
Device: aCRT ON — CRT device with AdaptivCRT enabled
  Arms: AdaptivCRT ON (aCRT ON, treatment group)
Device: aCRT OFF — CRT device with AdaptivCRT disabled
  Arms: AdaptivCRT OFF (aCRT OFF, control group)

SUMMARY:
The Mid-Q Response study is a prospective, multi-center, randomized controlled, interventional, single-blinded, post-market study.

The purpose of the Mid-Q Response study is to test the hypothesis that the AdaptivCRT (aCRT) algorithm is superior to standard CRT therapy regarding patient outcomes in CRT indicated patients with moderate QRS duration, preserved atrioventricular (AV) conduction and left bundle branch block (LBBB).

The study will be executed at approximately 60 centers in Asia. The subjects will be randomly assigned in a 1:1 ratio to the aCRT ON (Adaptive Bi-V and LV) group or the aCRT OFF (Nonadaptive CRT) group.

The primary objective is to test the hypothesis that aCRT ON increases the proportion of patients that improve on the Clinical Composite Score (CCS) compared to aCRT OFF at 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the study Informed Consent Form (ICF).
* Subject is indicated for a CRT device according to local guidelines.
* Subject has sinus rhythm at time of enrollment
* Subject has a moderately wide intrinsic QRS duration ≥120 ms and <150 ms
* Subject has Left Bundle Branch Block (LBBB) as documented on an ECG (preferably within 30 days prior to enrollment but up to 50 days is accepted) with Qs or rS in leads V1 and V2, and Mid-QRS notching or slurring in ≥2 of leads V1, V2, V5, V6, I, and aVL
* Subject has intrinsic, normal AV conduction as documented on an ECG by a PR interval ≤200 ms (preferably within 30 days prior to enrollment but up to 50 days is accepted).
* Subject has left ventricular ejection fraction ≤35% (documented within 180 days prior to enrollment).
* Subject has NYHA class II, III, or IV (documented within 30 days prior to enrollment) despite optimal medical therapy. Optimal medical therapy is defined as maximal tolerated dose of Beta-blockers and a therapeutic dose of ACE-I, ARB or MRA.

Exclusion Criteria:

* Subject is less than 18 years of age (or has not reached minimum age per local law if that is higher).
* Subject is not expected to remain available for at least 1 year of follow-up visits.
* Subjects has permanent atrial arrhythmias for which pharmacological therapy and/or cardioversion have been unsuccessful or have not been attempted.
* Subject is, or previously has been, receiving cardiac resynchronization therapy.
* Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Subject has unstable angina, or experienced an acute myocardial infarction (MI) or received coronary artery revascularization (CABG) or coronary angioplasty (PTCA) within 30 days prior to enrollment.
* Subject has a mechanical tricuspid heart valve or is scheduled to undergo valve repair or valve replacement during the course of the study.
* Subject is post heart transplant (subjects on the heart transplant list for the first time are not excluded).
* Subject has a limited life expectancy due to non-cardiac causes that would not allow completion of the study.
* Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to device implant).
* Subject meets any exclusion criteria required by local law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazutaka Aonuma, MD, Study Chair — University of Tsukuba Hospital
Locations (61):
- Gleneagles Jerudong Park Medical Centre, Bandar Seri Begawan, Brunei
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China
- Hong Kong (3):
  - Grantham Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia
- Japan (32):
  - University of Fukui Hospital, Fukui
  - Kokura Memorial Hospital, Fukuoka
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima Prefectural Hospital, Hiroshima
  - The Hospital of Hyogo College of Medicine, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Tokai University Hospital, Isehara
  - Kitasato University Hospital, Kanagawa
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Tohoku University Hospital, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki
  - University of Miyazaki Hospital, Miyazaki
  - Iwate Medical University Hospital, Morioka
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - The Sakakibara Heart Institute of Okayama, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
  - Sakurabashi Watanabe Hospital, Osaka
  - Japanese Red Cross Saitama Hospital, Saitama
  - Saitama Medical Center Jichi Medical University, Saitama
  - Saitama Medical University International Medical Center, Saitama
  - Shizuoka General Hospital, Shizuoka
  - Juntendo University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Yamagata Prefectural Central Hospital, Yamagata
  - Saiseikai Yokohama tobu Hospital, Yokohama
  - St. Marianna University Yokohama City Seibu Hospital, Yokohama
  - Oita University Hospital, Yufu
- Malaysia (5):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Serdang, Kajang
  - Sarawak Heart Center, Kota
  - Institut Jantung Negara - National Heart Institute, Kuala Lumpur
  - Sarawak Heart Centre, Kuching
- Makati Medical Center, Makati, Philippines
- Singapore (3):
  - Changi General Hospital, Singapore
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (9):
  - Sejong General Hospital, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (5):
  - National Taiwan University Hospital Hsin Chu Branch, Hsinchu
  - Kaohsing Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was multicentric and in a hospital setting, patients selected were heart failure patients in Asian countries indicated for CRT per local guidelines with moderately wide QRS (duration ≥120ms and <150ms), preserved AV conduction (PR interval ≤ 200 ms), along with a Left bundle branch block (LBBB).
Pre-assignment Details: Patients were enrolled as long as they met the inclusion criteria and were willing to consent. A total of 177 subjects were enrolled, of which 171 subjects were randomized between Adaptive and Conventional CRT.
Groups:
- AdaptivCRT ON (aCRT ON, Treatment Group): AdaptivCRT programmed to "Adaptive Bi-V and LV". The aCRT algorithm has been developed to provide RV-synchronized LV pacing when intrinsic AV conduction is normal or BiV pacing otherwise.
  aCRT ON: CRT device with AdaptivCRT enabled
- AdaptivCRT OFF (aCRT OFF, Control Group): AdaptivCRT programmed to "Nonadaptive CRT" (standard CRT). Control group subjects will be optimized per physician's discretion.
  aCRT OFF: CRT device with AdaptivCRT disabled
Period: Overall Study
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Started | 86 | 85
Completed | 80 | 78
Not Completed | 6 | 7
Not completed — Death | 5 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of subjects randomized following successful implant
Groups:
- Total: Total of all reporting groups
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group) | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (11.3) | 65.8 (13.7) | 66.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 57 | 60 | 117
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
NYHA class [Count of Participants; unit: Participants] — Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    NYHA class I | 1 | 1 | 2
    NYHA class II | 30 | 31 | 61
    NYHA class IIII | 52 | 47 | 99
    NYHA class IV | 3 | 6 | 9
LVEF [Mean (Standard Deviation); unit: percent] — Left ventricular ejection fraction
  percent | 27.0 (6.6) | 25.2 (6.5) | 26.1 (6.6)
QRS duration [Mean (Standard Deviation); unit: ms] | 136.9 (9.4) | 136.1 (9.0) | 136.5 (9.2)
PR interval [Mean (Standard Deviation); unit: ms] | 173.2 (21.0) | 174.3 (21.4) | 173.7 (21.1)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Composite Score
Description: The Clinical Composite Score (CCS) classifies patients according their clinical status at 6 months post-randomization into categories Improved, Unchanged, and Worsened. A patient is classified Worsened in case of death, hospitalization for worsening heart failure, worsened New York Heart Association (NYHA) class (using last observation carried forward), or worsened status on the Global Assessment Score. Also, patients that exit the study or cross over because of worsening heart failure are classified Worsened. A patient is classified Improved when not Worsened and there is an improvement in NYHA class or Global Assessment Score. Patients that are not Worsened or Improved are Unchanged including all patients that miss NYHA class and Global Assessment Score data and are not classified Worsened because of death, HF hospitalization, exit or crossover.
Time Frame: 6 months post-randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Number analyzed (Participants) | 86 | 85
Participants
  Improved | 66 | 68
  Unchanged | 10 | 11
  Worsened | 10 | 6
Statistical Analysis 1: Comparison: AdaptivCRT ON (aCRT ON, Treatment Group) vs AdaptivCRT OFF (aCRT OFF, Control Group); Test type: Superiority — Endpoint for statistical analysis is the proportion Improved; p = 0.61, Chi-squared

2. Secondary Outcome: Change in New York Heart Association (NYHA) Class
Description: NYHA class is an ordinal variable with higher classes indicating a worse degree of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: Baseline to 6 and 12 months post-randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Number analyzed (Participants) | 86 | 85
Participants
  Baseline: Class I | 1 | 1
  Baseline: Class II | 30 | 31
  Baseline: Class III/IV | 55 | 53
  Baseline: Not reported | 0 | 0
  3 Month: Class I | 24 | 22
  3 Month: Class II | 49 | 53
  3 Month: Class III/IV | 11 | 4
  3 Month: Not reported | 2 | 6
  6 Month: Class I | 23 | 27
  6 Month: Class II | 50 | 52
  6 Month: Class III/IV | 11 | 3
  6 Month: Not reported | 2 | 3
  12 Month: Class I | 35 | 32
  12 Month: Class II | 41 | 42
  12 Month: Class III/IV | 8 | 9
  12 Month: Not reported | 2 | 2
Statistical Analysis 1: Comparison: AdaptivCRT ON (aCRT ON, Treatment Group) vs AdaptivCRT OFF (aCRT OFF, Control Group); Due to limited number of subjects with NYHA class III or IV during follow-up, class III, IV, and death were grouped as a single category for analysis; Test type: Superiority; p = 0.63, Regression, Logistic; Proportional odds logistic regression model. Baseline NYHA class and time included as fixed covariates; Odds Ratio (OR) = 1.192, 95% CI 2-sided [0.579 to 2.455], Standard Error of Mean 0.367

3. Secondary Outcome: Occurrence of Hospitalizations for Worsening Heart Failure
Description: Defined as an event requiring inpatient hospitalization or invasive intervention
Time Frame: 12 months post-randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Number analyzed (Participants) | 86 | 85
Participants | 10 | 8
Statistical Analysis 1: Comparison: AdaptivCRT ON (aCRT ON, Treatment Group) vs AdaptivCRT OFF (aCRT OFF, Control Group); Test type: Superiority; p = 0.64, Regression, Cox; Adjusted for NYHA class and sex; Hazard Ratio (HR) = 1.250, 95% CI 2-sided [0.492 to 3.175], Standard Error of Mean 0.476

4. Secondary Outcome: All-cause Mortality
Description: All-cause mortality in the aCRT ON group vs the aCRT OFF group
Time Frame: 12 months post-randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Number analyzed (Participants) | 86 | 85
Participants | 5 | 6
Statistical Analysis 1: Comparison: AdaptivCRT ON (aCRT ON, Treatment Group) vs AdaptivCRT OFF (aCRT OFF, Control Group); Test type: Superiority; p = 0.78, Log Rank

5. Secondary Outcome: Cardiovascular-related Mortality
Description: Defined as all cardiac deaths as well as any cardiovascular deaths that are not directly a result of mechanical or electrical heart dysfunction.
Time Frame: 12 months post-randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
Number analyzed (Participants) | 86 | 85
Participants | 3 | 3
Statistical Analysis 1: Comparison: AdaptivCRT ON (aCRT ON, Treatment Group) vs AdaptivCRT OFF (aCRT OFF, Control Group); Test type: Superiority; p = 0.98, Regression, Cox; Hazard Ratio (HR) = 1.020, 95% CI 2-sided [0.206 to 5.056], Standard Error of Mean 0.817

ADVERSE EVENTS:
Time Frame: The data were collected from the time the subject signed informed consent until they completed the study, 12 months post-randomization.
Description: All serious, cardiovascular, device or procedure-related events were considered reportable. Pre-existing conditions that existed prior to study participation were not considered reportable, unless the condition recurred after the patient had recovered from the pre-existing condition, or the condition worsened in intensity or frequency during the study. Planned hospitalizations for a pre-existing condition without serious deterioration in health were not considered SAEs.
Arm/Group | AdaptivCRT ON (aCRT ON, Treatment Group) | AdaptivCRT OFF (aCRT OFF, Control Group)
All-Cause Mortality (participants affected / at risk) | 5/86 | 6/85
Serious Adverse Events (participants affected / at risk) | 27/86 | 24/85
Other Adverse Events (participants affected / at risk) | 8/86 | 14/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdaptivCRT ON (aCRT ON, Treatment Group) (N=86) | AdaptivCRT OFF (aCRT OFF, Control Group) (N=85)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 7 (7) | 7 (12)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 0 (0) | 1 (1)
Medical device site inflammation (General disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdaptivCRT ON (aCRT ON, Treatment Group) (N=86) | AdaptivCRT OFF (aCRT OFF, Control Group) (N=85)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Device stimulation issue (Product Issues) | 3 (3) | 7 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04180696/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04180696/SAP_001.pdf